CLINICAL TRIAL: NCT06489860
Title: SARS-CoV-2 Safety Study for the Treatment of COVID-19
Acronym: SARS-CoV-2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: My record is not overseen by an IRB, I change the Overall Status to Withdrawn.
Sponsor: DHA Coffee Co., Ltd (Industry)
Responsible Party: Principal Investigator, Do Van Tin, DHA Coffee Co., Ltd, DHA Coffee Co., Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHACoffee
Record Dates: First submitted 2024-03-05; First posted 2024-07-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Intervention Model Description: SARS-CoV-2. Directions: For adults and for Children 1-12 years old. Indication: SARS-CoV-2.
  Ingredient: Organic Rice 95% and Honey 5% Powder (whole) 1g.
Masking Description: Directions: For adults and for Children 1-12 years old. Indication: SARS-CoV-2 Ingredient: Organic Rice 95% and Honey 5% Powder (whole) 1g. Mix one packet with 6.8 fl oz (200 ml) of hot water (220ºF/100ºC) about three minutes until dissolved.
  Participants: Use 4 to 5 packets, use one pack each time after two hours. Humidification: <5% Dosage Form: Powder form Dosage Strength: 1.0 G/ 1 Unit, use one pack of 1 g for each time Use within two years from the manufacturing date. Storage normal conditions in dry, cool and temperature from 15 °C to 32 °C Store in a dry environment (75% humidity).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARS-CoV-2 Safety Study for the Treatment of COVID-19 (Experimental): Directions: For adults and for Children 1-12 years old. Indication:SARS-CoV-2 Ingredients: Organic Rice 95% and Honey 5% Powder (whole) 1g. Mix one packet with 6.8 fl oz (200 ml) of hot water (220ºF/100ºC) about three minutes until dissolved.
  Participants: Use 4 to 5 packets, use one pack each time after two hours. Humidification: <5% Dosage Form: Powder form Dosage Strength: 1.0 G/ 1 Unit, use one pack of 1 g for each time Use within two years from the manufacturing date. Storage normal conditions in dry, cool and temperature from 15 °C to 32 °C Store in a dry environment (75% humidity).
  Interventions: Drug: HIV; Drug: Malignant Neoplasms Safety Study for the Treatment of Neoplasms

INTERVENTIONS:
Drug: HIV — Directions: For adults and for Children 1-12 years old. Indication: HIV Ingredient: Organic Rice 93% and Honey 7% Powder (whole) 1g. Masking: None (Open Label) Mix one packet with 6.8 fl oz (200 ml) of hot water (220ºF/100ºC) about three minutes until dissolved. Participants: Use 4 to 5 packets, use one pack each time after two hours.
  Humidification: <5% Dosage Form:
  Powder form Dosage Strength: 1.0 G/ 1 Unit, use one pack of 1 g for each time Use within two years from the manufacturing date
  Other Names: HIV Safety Study for the Treatment of Anti-AIDS Drug
Drug: Malignant Neoplasms Safety Study for the Treatment of Neoplasms — Directions: For adults and for Children 1-12 years old. Indication: Malignant Neoplasms . Ingredient: Organic Rice 92% and Honey 8% Powder (whole) 1g. Mix one packet with 6.8 fl oz (200 ml) of hot water (220ºF/100ºC) about three minutes until dissolved. Participants: Use 4 to 5 packets, use one pack each time after two hours. Humidification: <5% Dosage Form: Powder form Dosage Strength: 1.0 G/ 1 Unit, use one pack of 1 g for each time Use within two years from the manufacturing date.
  Other Names: Malignant Neoplasms

SUMMARY:
SARS-CoV-2 produced strong pluripotent stem cells and brain cells to protect Telomere chromosomes to maintain Acid Deoxyribonucleic (ADN) Molecules.

DETAILED DESCRIPTION:
SARS-CoV-2 produced strong pluripotent stem cells and brain cells to change and disappear defective cells in virus variants, Covid-19 disease. Pluripotent stem cells produced strong cells serve as a repair system, replacing damaged cells, defective cells and dead cells.

CHEMISTRY:

SARS-CoV-2 does not use any chemicals, no colors and no additives and no preservatives.

Toxicology:

SARS-CoV-2 product is not adverse effect, non-toxic and no pharmacal toxicology.

SARS-CoV-2 is not placebo drug

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2

Exclusion Criteria:

Ages: 1 Year to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Directions: For adults and for Children 1-12 years old.
Enrollment: 0 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-04 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 | From September to October, 2024
  1. Parameters: Humidification, Unit: %, Result: 4.40, Test Method: ISO 7932: 2004.
  2. Cadmium (Cd), mg/Kg, 0.1, CASE.TN.0018 (Ref. AOAC 999.11).
  3. Hydrargyrum (Hg), mg/Kg, 0.01, CASE.TN.0141 (Ref . EPA Method 7473).
  4. Plumbum (Pb), mg/liter, 0.001, SMEWW3030E 2017: 31258: 2017.
  5. Cadmium (Cd), mg/liter, 0.0001, SMEWW3030E 2017: 31258: 2017. .
  6. Arsen (As), mg/liter, 0.001, SMEWW3030E 2017: 31258: 2017.
  7. Hydrargyrum (Hg), mg/liter, 0.0001, SMEWW3030E 2017: 31258: 2017.
  8. Clostridium perfringents, CFU/g, < 10, ISO 7937:2004.
  9. Coliforms, CFU/g, < 10, ISO 4832:2006 (*).
  10. Escherichia coli, CFU/g, < 10, ISO 7937:2006.
  11. Salmonella, /25g, Not detected, ISO 7937:2007.
  12. Staphylococcus aureus, CFU/g, < 10, ISO 7937:2008.
  13. Total Yeasts molds, CFU/g, < 10, ISO 7937:2009.
  14. Total Aerobic Microbial, CFU/g, 1.0 x 100, ISO 7937:2010.
  15. Vibrio parahaemolyticuc, /25g, Not detected, ISO 7937:2011. .

CONTACTS AND LOCATIONS:
Overall Officials: PHUOC T DO, Principal Investigator — DHA Coffee Co., Ltd

IPD SHARING:
Plan to Share IPD: No
20 -1 g Packets Net Weight 0.70 oz (20 g) Directions: For adults and for Children 1-12 years old. Indication: Treated the SARS-CoV-2 treatment COVID-19 within 20 days Ingredient: Organic Rice 95% and Honey 5% Powder (whole) 1g. Mix one packet with 6.8 fl oz (200 ml) of hot water (220ºF/100ºC) about three minutes until dissolved.
  Participants: Use 4 to 5 packets, use one pack each time after two hours. Use within two years from the manufacturing date. Humidification: <5% Dosage Form: Powder form Dosage Strength: 1.0 G/ 1 Unit, use one pack of 1 g for each time Storage normal conditions in dry, cool and temperature from 15 °C to 32 °C Store in a dry environment (75% humidity).

REFERENCES:
- [Result] Zarin DA, Tse T, Williams RJ, Califf RM, Ide NC. The ClinicalTrials.gov results database--update and key issues. N Engl J Med. 2011 Mar 3;364(9):852-60. doi: 10.1056/NEJMsa1012065. PMID 21366476
- See also: This Website was pause hosting website — http://dhacoffee.com